CLINICAL TRIAL: NCT00075166
Title: A Prospective, Randomized Trial Comparing Surgery Versus Radiosurgery for the Treatment of Metastatic Brain Tumors
Brief Title: Surgery Versus Radiosurgery to Treat Metastatic Brain Tumors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040066; 04-N-0066
Record Dates: First submitted 2004-01-02; First posted 2004-01-05 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Brain Neoplasms; Neoplasm Metastasis
Keywords: Stereotactic; Carcinoma; Melanoma; Surgical Resection; Metastases; Metastatic Brain Tumor; Surgery; Radiosurgery; Treatment
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis; Carcinoma; Melanoma | interventions — Craniotomy

INTERVENTIONS:
Procedure: Stereotactic surgery (SRS)
Procedure: Craniotomy

SUMMARY:
This study will compare the effectiveness of craniotomy to that of stereotactic surgery (SRS) for the treatment of metastatic brain tumors - tumors that first develop elsewhere in the body and then travel to the brain. Craniotomy is surgical removal of the tumors through an operation. SRS consists of highly focused radiation doses to the tumors. Neither treatment is experimental and both have shown benefits to patients with metastatic brain tumors. This study will determine whether one treatment is superior to the other in prolonging patient survival.

Patients 21 years of age and older with one to three metastatic brain tumors may be eligible for this study. Participants will have a medical history and physical examination, blood and urine tests, an electrocardiogram, and chest x-ray. They will then be randomly assigned to undergo either surgery or SRS. Before either procedure, patients will have a magnetic resonance imaging (MRI) scan. MRI uses a strong magnetic field and radio waves to obtain images of the brain. Patients scheduled for SRS will have a computed tomography (CT) scan in addition to the MRI. CT uses X-rays to obtain images of the brain. During the CT, a contrast agent is injected through an IV tube placed in a vein to enhance the CT images. For both the MRI and CT tests, the patient lies on a table that slides into a cylindrical scanner. The MRI usually lasts between 45 and 90 minutes, while the CT scan lasts for about 30 to 60 minutes.

Patients scheduled for surgery will have general anesthesia or local anesthesia with sedation. They will be in intensive care after the surgery until their condition is stable. Before being discharged home, they will have another MRI scan. The surgical sutures or staples will be removed 7 to 10 days after surgery.

Patients scheduled for SRS will have their scalp numbed with medicine and their head will be placed in a head frame. A CT scan will be done on the morning of the procedure to plan the treatment. Around noon, the treatment, which consists of brief exposures to radiation, will be administered with the patient positioned comfortably on a treatment couch. The treatment will be completed in 1 to 2 hours, after which the head frame will be removed. After a brief period of observation, the patient will be discharged home.

Patients will return to NIH for follow-up visits within 4 weeks after surgery or SRS and then every 3 months after that for a medical history, physical examination, and MRI scan, and to complete a quality of life questionnaire.

DETAILED DESCRIPTION:
Introduction: Metastatic brain tumors occur more frequently than primary brain tumors and occur in approximately 25% of patients who die of cancer each year. The main treatment goals for patients with brain metastases are the relief of neurological symptoms and long-term control of the tumors. Glucocorticoids and external beam whole brain radiation therapy (WBRT) comprise the current standard of care and increase median survival from one month to three to six months. Patients with three or less tumors (greater than 70% of patients) also commonly undergo surgery or stereotactic radiosurgery (SRS) with the goal of lengthening survival. Two prospective randomized trials have shown a significant survival benefit for patients undergoing surgical resection of single tumors in combination with WBRT compared to patients receiving WBRT alone. Although there have been no prospective randomized studies comparing SRS and WBRT to WBRT alone, there have been numerous large retrospective series reporting a significant survival benefit from SRS. To date, a prospective randomized trial comparing surgery to SRS has not been reported. Despite the lack of rigorous data, there are proponents for each of these treatment modalities. Those in favor of surgery cite the ability to achieve a complete resection in most cases, the almost immediate relief of symptoms, and the low rate of local recurrence. Those in favor of SRS cite an equivalent degree of local tumor control compared to surgery, the relative ease of the one day outpatient procedure, and the ability to treat lesions in deeper brain structures.

Objectives: We plan to determine in a prospective randomized manner if surgery is superior to SRS for prolonging survival in patients with one to three surgically accessible brain tumors.

Study Population: Patients aged twenty one years and older with one to three brain metastases will be assessed for enrollment in this study.

Design: Patients who meet eligibility criteria will be randomly assigned to undergo either surgery or SRS for their tumors. Patients will then be followed at regularly scheduled intervals for the duration of their disease.

Outcome measures: The primary outcome measure will be time of survival following treatment. Among the secondary outcomes that will be measured over time are tumor recurrence or progression, neurologic sign or symptom development, functional independence, steroid and anticonvulsant use, and overall quality of life.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must:

1. be 21 years of age or older.
2. have a histologically confirmed primary malignancy.
3. be able to undergo an MRI scan of the brain.
4. have one to three intraparenchymal brain metastases as identified on a brain MRI scan with intravenous contrast.
5. have contrast enhancing tumor(s) that are well circumscribed and less than or equal to 4.0 cm in any dimension.
6. be appropriate for either procedure as determined by both a neurosurgeon and a radiation oncologist.

EXCLUSION CRITERIA:

Patients must not:

1. have tumor(s) in the midbrain, pons, or medulla - patients undergoing surgical resections in these areas are highly likely to develop significant neurological deficits or death.
2. have tumors within 10 millimeters of the optic apparatus (nerves and chiasm) or the area postrema - patients undergoing SRS to these areas are at significant risk of developing permanent blindness or intractable nausea.
3. be poor operative candidates from an anesthetic point of view secondary to other major medical illnesses - the risk of undergoing general anesthesia outweighs the potential benefit of undergoing surgical resection of a brain metastasis.
4. have a coagulopathy demonstrated by an abnormal prothrombin time, activated partial thromboplastin time, or thrombocytopenia (platelet count less that 150,000 platelets/mm3) - the risk of developing uncontrollable intra-operatively bleeding outweighs the potential benefit of undergoing surgical resection of a brain metastasis.
5. have radiographic or cerebrospinal fluid specimen evidence of widespread leptomeningeal metastasis - neither surgery nor SRS is a useful treatment modality for this condition.
6. significant psychiatric impairments which, in the opinion of the investigators, will interfere with the proper administration or completion of the protocol - self explanatory.
7. acute or untreated infections (viral, bacterial or fungal) - patients with active infections are highly likely to have spread of their infections to the brain as a result of a craniotomy.
8. be pregnant at the time of the randomized treatment - general anesthesia and surgery may subject the fetus to unacceptable risks. Also, the NIH does not offer full obstetrical services in the event that medical care to the mother and/or fetus is required. Pregnant women presenting with brain metastases will be referred to facilities offering OB/GYN services.
9. be prisoners or other institutionalized individuals - these individuals are at risk of being susceptible to undue influences to participate in a research protocol against their free will.
10. have a diagnosis of germ cell tumor, lymphoma or small cell lung cancer - these tumors are highly radiosensitive and should therefore be treated with radiation.
11. have any of the following: aneurysm clip, implanted neural stimulator, implanted cardiac pacemaker or auto defibrillator, cochlear implant, ocular foreign body or implant [e.g. metal shavings, retinal clips], or insulin pump as these items would be contra-indications to undergoing an MRI scan.
12. have an allergy to iodine or shellfish or have previously had an allergic reaction to iodinated-contrast agents as this is a contra-indication to undergoing a contrast enhanced CT of the brain - a contrast enhanced CT of the brain is required for the planning of SRS.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 2003-12; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Wen PY, Loeffler JS. Brain metastases. Curr Treat Options Oncol. 2000 Dec;1(5):447-58. doi: 10.1007/s11864-000-0072-3. PMID 12057152
- [Background] Johnson JD, Young B. Demographics of brain metastasis. Neurosurg Clin N Am. 1996 Jul;7(3):337-44. PMID 8823767
- [Background] Posner JB. Management of brain metastases. Rev Neurol (Paris). 1992;148(6-7):477-87. PMID 1448668